CLINICAL TRIAL: NCT06650358
Title: CLINICAL OUTCOMES of BILATERAL PSEUDOPHAKIC PATIENTS with a LIGHT ADJUSTABLE LENS+ (LAL)+ IMPLANTED in AT LEAST ONE EYE
Brief Title: Clinical Outcomes of Patients with LAL+ in At Least One Eye
Status: Enrolling by invitation | Type: Observational
Sponsor: Frank A. Bucci, Jr., M.D. (Other)
Responsible Party: Sponsor-Investigator, Frank A. Bucci, Jr., M.D., Medical Director, Bucci Laser Vision Institute
Organization: Bucci Laser Vision Institute (Other)
Other Study IDs: IIT-004-02
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: IOL, Cataract
Keywords: LAL+; Light Adjustable Lens+; Mix and match IOLs
MeSH Terms: conditions — Intraocular Lymphoma; Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- LAL+: Bilateral pesudophakic adults implanted with the LAL+ in at least one eye
  Interventions: Device: Light Adjustable Lens+

INTERVENTIONS:
Device: Light Adjustable Lens+ — The Light Adjustable Lens+ (LAL+) is a posterior chamber, UV absorbing, three-piece, foldable, photo reactive silicone intraocular lens with a squared-posterior optic edge intended to be implanted in the capsular bag following phacoemulsification. Selective exposure to the implanted LAL+ using the Light Delivery Device (LDD) to deliver a spatially profiled UV light produces modifications in the lens curvature resulting in a spherical or spherocylindrical power change postoperatively. A subsequent lock-in exposure is delivered to the implanted LAL+ to stabilize the lens power. The LAL+ has a modified aspheric anterior surface that creates a small continuous increase in central lens power, which is designed to slightly extend the depth of focus.

SUMMARY:
The objective of this study is to collect data on bilateral pseudophakic patients implanted with the RxSight Light Adjustable Lens+ (LAL+) in at least one eye

DETAILED DESCRIPTION:
A retrospective-prospective, single-center study will be conducted. Patient charts will be retrospectively reviewed to collect data from the patient's comprehensive preoperative exam. Subjects will attend one stud visit post final LDD light treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults with bilateral pseudophakia who have been implanted with the LAL+ in at least one eye and who have completed LDD light treatments
* Sign a written Informed Consent Form

Exclusion Criteria:

* Visually significant eye disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: PI's current patients
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction | 3-18 months after phacoemulsification
  Description: Subjective questionnaire explores the frequency/need for glasses for various visual functions at distance/intermediate/near, experience with dysphotopsias, and overall satisfaction of visual function without glasses.

CONTACTS AND LOCATIONS:
Locations (1):
- Bucci Laser Vision Institute, Wilkes-Barre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No